CLINICAL TRIAL: NCT04519476
Title: A Pilot Study Examining Selinexor's Ability to Overcome Resistance in Multiple Myeloma Patients Who Are Refractory to Lenalidomide-containing Therapy.
Brief Title: Selinexor Treatment for Multiple Myeloma Patients Who Are Refractory to Lenalidomide-containing Therapy.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oncotherapeutics (Industry)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-321
Record Dates: First submitted 2020-08-12; First posted 2020-08-19 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Refractory Multiple Myeloma
Keywords: Selinexor; Lenalidomide-Refractory; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor; Lenalidomide; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: A pilot study examining selinexor's ability to overcome resistance in multiple myeloma patients who are refractory to lenalidomide-containing therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Selinexor/Lenalidomide/Steroids (Experimental): All subjects enrolled will receive: 1) selinexor, PO, at 60 mg once weekly on days 1-28 of a 28-day cycle, 2) lenalidomide, PO, 10 mg daily on days 1-21 of 28-days cycle and 3) methylprednisolone at the same dose and schedule as the last lenalidomide-containing regimen if it contained steroids. If patient's qualifying lenalidomide-containing regimen contained different type of steroid (e.g. prednisone, dexamethasone, etc.) then patient on this study will receive methylprednisolone at the equivalent dose and schedule.
  Interventions: Drug: Selinexor; Drug: Lenalidomide; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Selinexor — Selinexor (KPT-330) is a first-in-class, oral selective exportin 1 (XPO1) inhibitor (1,2). Selinexor functions by binding with and inhibiting the nuclear export protein XPO1 (also called CRM1), leading to the accumulation of tumor suppressor proteins in the cell nucleus along with inhibition of translation of oncoprotein mRNAs.
  Other Names: KPT-330
Drug: Lenalidomide — Immunomodulatory drug
  Other Names: Revlimid
Drug: Methylprednisolone — Glucocorticoid, steroid
  Other Names: Medrol

SUMMARY:
This is a pilot study evaluating the safety and efficacy of selinexor among multiple myeloma (MM) patients that are refractory to lenalidomide-containing regimens with or without steroids.

DETAILED DESCRIPTION:
This is a pilot, multi-center, open-label study evaluating selinexor's ability to overcome resistance for multiple myeloma patients who are refractory to lenalidomide-containing therapies.

Enrollment:

The study will enroll up to a total of 22 Multiple Myeloma (MM) patients with progressive disease.

Study Assessments:

The study will consist of:

1. screening period;
2. study treatment until disease progression or intolerable toxicity;
3. a final assessment to occur up to 28 days after the end of the last treatment cycle; and
4. follow-up period.

The screening period will be conducted within 14 days before baseline (baseline being day 1 of cycle 1, before study drug administration). During this period, a medical history will be obtained along with complete physical examination including vital signs measurements, height, weight, Eastern Cooperative Oncology Group (ECOG) performance status, and 12-lead electrocardiogram (EKG). MM assessments will be performed, including β2 microglobulin (β2M), serum free light chain (SFLC) serum and urine protein electrophoresis, quantification of serum immunoglobulins, urine and serum immunofixation, and 24-hour total protein. An additional serum sample will be obtained for evaluation of biomarkers. In addition, a postero-anterior and lateral chest radiographs, skeletal survey, and a bone marrow aspirate (BM) and biopsy will be performed within 28 days of baseline. Clinical laboratory tests including hematology, clinical chemistry (blood urea nitrogen [BUN], serum creatinine, uric acid, lactate dehydrogenase [LDH], total bilirubin, alkaline phosphatase, aspartate aminotransferase [AST] and alanine aminotransferase [ALT]), electrolytes (potassium, sodium, chloride and calcium), random glucose, total protein, amylase, albumin, and urinalysis as well as serum pregnancy tests for females of child-bearing potential (FCBPs). Subjects will also be asked to fill out quality of life assessments at several time points during this study.

Subjects eligible for this study will receive treatment with study drug until disease progression or intolerable toxicity does not allow ongoing treatment.

Assessments:

Schedule of assessments: Subjects that meet the inclusion/exclusion criteria during the screening period will continue to Day 1 of Cycle 1, when baseline evaluations will be conducted. Subjects who continue to meet the inclusion/exclusion criteria will be enrolled in the trial and study drug will be administered. During Cycle 1, subjects will also have study visits during which assessments will be performed on Days 8, 15 and 22. MM assessments will be performed on Day 22 during all subsequent cycles. Starting with Cycle 2, study visits will take place on Days 1 and 22. See Table 1

Assessment overview: During the treatment period, each subject will have clinical laboratory tests performed to monitor for potential toxicity. Additional procedures performed at these visits will include monitoring for adverse events (AEs), review of concomitant medications and other support therapies (e.g. growth factors and transfusion), MM disease assessments, ECOG performance status, vital signs measurements, and physical examination. Subjects will remain on study until documentation of progressive disease (PD) as defined by the International Myeloma Working Group (IMWG) criteria. Subjects with stable disease will remain in the study. For subjects who show disappearance of urine and serum M-protein by protein electrophoresis and immunofixation on 2 consecutive assessments and the subject shows no other signs of disease activity, a bone marrow (BM) aspirate and biopsy will be required to confirm their CR. A BM aspirate and biopsy will not be required for subjects in any other response group categories.

Up to twenty-eight days after the last dose of study drug, subjects are to complete a final assessment (herein referred to as the End-of-Study treatment visit). Procedures to be conducted at this visit include a MM disease assessment, measurement of vital signs and weight, a complete physical examination, assessment of adverse events, a review of concomitant medications, assessment of ECOG performance status, hematology and clinical chemistry laboratory tests including electrolytes, total protein, amylase and albumin, and an assessment of response to treatment with the use of SFLC assay and ratio, serum and urine protein electrophoresis, quantification of serum immunoglobulins, urine and serum immunofixation, 24-hour total urine protein, and serum β2M. Subjects who withdraw from the study before the completion of the eight 28-day cycle evaluation periods will have all End- of-Study treatment assessments performed at their final visit.

Following the End-of-Study treatment visit, subjects will be monitored for PD and survival by clinic visits every 3 months and every 6 months, respectively, until alternate therapy needs to be started or death intervenes.

Dosing Regimens:

All subjects enrolled will receive (Dose Level 0) 1) selinexor, PO, at 60 mg once weekly on days 1, 8, 15, and 22 of a 28-days cycle, 2) lenalidomide, PO, 10 mg daily on days 1-21 of a 28-day cycle and 3) steroids at the same dose and schedule as the last lenalidomide-containing regimen if it contained steroids that they had failed to meet eligibility for this study.

Recommended Concomitant Therapy:

Subjects may receive full supportive care, including hydration prophylaxis, treatment with a 5-HT3 antagonist and/or other anti-nausea agents, antibiotics, antivirals, vitamins, and supplements as appropriate. Patients should receive anti-platelet therapy with baby aspirin or other agents if they have additional risk factors for developing thrombotic events.

Number of Patients (planned): 22

Study Population: Multiple myeloma patients who are refractory to a lenalidomide-containing therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible to enroll in this study:

  1. Age ≥ 18 year of age.
  2. Willing and able to provide written informed consent in accordance with federal, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure.
  3. Able to adhere to the study visit schedule and other protocol requirements.
  4. ECOG Performance Status (PS) of ≤ 2.
  5. Has a diagnosis of MM based on standard criteria (9) as follows:

Major criteria:

1. Plasmacytomas on tissue biopsy.
2. Bone marrow plasmacytosis (greater than 30% plasma cells).
3. Monoclonal immunoglobulin spike on serum electrophoresis IgG greater than 3.5 g/dL or IgA greater than 2.0 g/dL or kappa or lambda light chain excretion greater than 1 g/day on 24-hour urine protein electrophoresis.

Minor criteria:

1. Bone marrow plasmacytosis (10% to 30% plasma cells).
2. Monoclonal immunoglobulin present but of lesser magnitude than given under major criteria.
3. Lytic bone lesions.
4. Normal IgM less than 50 mg/dL, IgA less than 100 mg/dL, or IgG less than 600 mg/dL.

   Any of the following sets of criteria will confirm the diagnosis of multiple myeloma:

   • any 2 of the major criteria

   • major criterion 1 plus minor criterion 2, 3, or 4

   • major criterion 3 plus minor criterion 1 or 3

   • minor criteria 1, 2, and 3, or 1, 2, and 4

6. Currently has MM with measurable disease, defined as:

* a monoclonal immunoglobulin spike on serum electrophoresis of at least 0.5 g/dL and/or
* urine monoclonal protein levels of at least 200 mg/24 hours
* for patients without measurable serum and urine M-protein levels, an involved SFLC > 100 mg/L or abnormal SFLC ratio 7. Currently has progressive MM: MM patients that are relapsed or have refractory disease from at least 3 regimens or lines of therapy are eligible for enrollment provided they fulfill the other eligibility criteria:
* patients are considered relapsed, when they progress greater than 8 weeks from their last dose of treatment
* patients are refractory when they progress while currently receiving the treatment or within 8 weeks of its last dose 8. Previous exposure to lenalidomide: failed lenalidomide (> 10 mg)-containing regimen (lenalidomide- containing regimen could be any prior regimen and is not required to be a part of their most recent treatment) and have received a proteasome inhibitor, an immunomodulatory agent and an anti-CD38 antibody therapy.

  9. Adequate hepatic function within 28 days prior to C1D1: Total bilirubin < 1.5 × upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 × ULN), and Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) normal to < 2 × ULN.

  10. Adequate renal function within 28 days prior to C1D1 as determined by serum creatinine of ≤1.5 mg/dL OR estimated CrCl of > 60 mL/min, calculated using the Cockcroft and Gault formula (140 - Age) • Mass (kg)/ (72 • creatinine mg/dL); multiply by 0.85 if female (10)(Appendix 5).

  11. Adequate hematopoietic function within 7 days prior to C1D1: total WBC count ≥1500/mm3, ANC ≥1000/mm3, hemoglobin ≥8.5 g/dL and platelet count ≥75,000/mm3 (patients for whom <50% of BM nucleated cells are plasma cells) or ≥50,000/mm3 (patients for whom ≥50% of BM nucleated cells are plasma cells).

  12. Patients receiving hematopoietic growth factor support, including erythropoietin, darbepoetin, G-CSF, GM-CSF, and platelet stimulators (e.g., eltrombopag, romiplostim, or interleukin-11) must have a 2-week interval between growth factor support and the Screening assessments, but they may receive growth factor support during the study.

  13. Patients must have:
* At least a 2-week interval from the last red blood cell (RBC) transfusion prior to the start of study treatment
* At least a 1-week interval from the last platelet transfusion prior to the start of study treatment
* However, patients may receive RBC and/or platelet transfusions as clinically indicated per institutional guidelines during the study 14. Patients must be registered into the mandatory REVLIMID REMS™ program and be willing and able to comply with the requirements of the REVLIMID REMS™ program.

  15. Female patients of childbearing potential (FCBP) must have a negative serum pregnancy test at Screening. Female patients of childbearing potential and fertile male patients who are sexually active with a female of childbearing potential must use highly effective methods of contraception throughout the study and for 3 months following the last dose of study treatment, specifically:
* FCBP† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting treatment and must either commit to continued abstinence from heterosexual intercourse or use acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, and at least 28 days before she starts therapy. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.

  * A FCBP (female of childbearing potential) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months) Able to take aspirin (acetylsalicylic acid, ASA) at 81 or 325 mg/daily as antiplatelet therapy if platelet count is above 30 x 109/L (subjects intolerant to ASA may use warfarin or low molecular weight heparin)

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria are not eligible to enroll in this study:

  1. Has received selinexor or another XPO1 inhibitor previously.
  2. Prior malignancy that required treatment or has shown evidence of recurrence (except for non-melanoma skin cancer or adequately treated cervical carcinoma in situ) during the 5 years prior to randomization. Cancer treated with curative intent for >5 years previously and without evidence of recurrence will be allowed.
  3. Has any concurrent medical condition or disease (e.g., uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection, POEMS syndrome [polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes], primary amyloidosis, etc.) that is likely to interfere with study procedures.
  4. Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to Cycle 1 Day 1 (C1D1). Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are acceptable.
  5. Known intolerance, hypersensitivity, or contraindication to glucocorticoids.
  6. Known hypersensitivity to compounds of similar chemical or biological composition to thalidomide and lenalidomide or steroids.
  7. Concurrent use of other anti-cancer agents or treatments.
  8. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
  9. Severe hypercalcemia, i.e., serum calcium ≥ 12 mg/dL (3.0 mmol/L) corrected for albumin
  10. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
  11. Pregnant or breastfeeding females.
  12. BSA <1.4 m2 at baseline, calculated by the Dubois (58) or Mosteller (59) method.
  13. Life expectancy of less than 3 months.
  14. Major surgery within 4 weeks prior to C1D1.
  15. Active, unstable cardiovascular function, as indicated by the presence of:

  1. Symptomatic ischemia, or 2. Uncontrolled clinically significant conduction abnormalities (e.g., patients with ventricular tachycardia on anti-arrhythmic are excluded; patients with first degree atrioventricular block or asymptomatic left anterior fascicular block/right bundle branch block will not be excluded), or 3. CHF of New York Heart Association Class ≥3 or known left ventricular ejection fraction < 40%, or 4. MI within 3 months prior to C1D1. 16. Known active HIV infection or HIV seropositivity. 17. Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus ribonucleic acid (RNA) or hepatitis B virus surface antigen.

  18. Any active GI dysfunction interfering with the patient's ability to swallow tablets, or any active GI dysfunction that could interfere with absorption of study treatment.

  19. Inability or unwillingness to take supportive medications such as anti-nausea and anti-anorexia agents as recommended by the National Comprehensive Cancer Network® (NCCN) Clinical Practice Guidelines in Oncology (CPGO) (NCCN CPGO) for antiemesis and anorexia/cachexia (palliative care).

  20. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.

  21. Contraindication to any of the required concomitant drugs or supportive treatments.

  22. Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12-29 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Overall Response | 30 months
  Overall Response Rate ([ORR]=CR +VGPR+ PR)
Clinical Benefit Rate | 30 months
  Clinical Benefit Rate ([CBR]= CR+VGPR+PR+MR)

SECONDARY OUTCOMES:
Adverse Events Occurrences | 30 months
  Occurrence of adverse events throughout the study, graded via CTCAE v.5.0
Time to progression (TTP) | 30 months
  defined as the time from the initiation of therapy to progressive disease
Progression-free survival (PFS) | 30 months
  defined as the time from initiation of therapy to progressive disease or death from any cause, whichever occurs first
Time to first response | 30 months
  defined as the time from the initiation of therapy to the first evidence of confirmed clinical benefit defined as > minimal response (MR, including patients who achieved a complete response (CR), very good partial response (VGPR), partial response (PR), or MR
Duration of Response (DOR) | 30 months
  defined as the time from the first response to progressive disease
Overall survival (OS) | 30 months
  defined as the time from initiation of therapy to death from any cause or last follow-up visit

OTHER OUTCOMES:
Measuring levels of multiple myeloma specific biomarkers such as M-Protein and BCMA | 30 months; duration of each cycle in this study is 28 days
  Levels will be measure on Day 1 Cycle 1 (baseline), Day 8 Cycle 1, Day 15 Cycle 1, Day 22 Cycle 1, and on Day 22 of every cycle thereafter. Duration of each cycle in this study is 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: James R Berenson, MD, Principal Investigator — Oncotherapeutics
Locations (1):
- James R Berenson, MD, Inc., West Hollywood, California, United States

IPD SHARING:
Plan to Share IPD: No
We will share overall demographics of the study population, clinical responses, AEs and SAEs.

REFERENCES:
- [Background] Abdul Razak AR, Mau-Soerensen M, Gabrail NY, Gerecitano JF, Shields AF, Unger TJ, Saint-Martin JR, Carlson R, Landesman Y, McCauley D, Rashal T, Lassen U, Kim R, Stayner LA, Mirza MR, Kauffman M, Shacham S, Mahipal A. First-in-Class, First-in-Human Phase I Study of Selinexor, a Selective Inhibitor of Nuclear Export, in Patients With Advanced Solid Tumors. J Clin Oncol. 2016 Dec;34(34):4142-4150. doi: 10.1200/JCO.2015.65.3949. Epub 2016 Oct 31. PMID 26926685
- [Background] Gounder MM, Zer A, Tap WD, Salah S, Dickson MA, Gupta AA, Keohan ML, Loong HH, D'Angelo SP, Baker S, Condy M, Nyquist-Schultz K, Tanner L, Erinjeri JP, Jasmine FH, Friedlander S, Carlson R, Unger TJ, Saint-Martin JR, Rashal T, Ellis J, Kauffman M, Shacham S, Schwartz GK, Abdul Razak AR. Phase IB Study of Selinexor, a First-in-Class Inhibitor of Nuclear Export, in Patients With Advanced Refractory Bone or Soft Tissue Sarcoma. J Clin Oncol. 2016 Sep 10;34(26):3166-74. doi: 10.1200/JCO.2016.67.6346. Epub 2016 Jul 25. PMID 27458288